CLINICAL TRIAL: NCT00816244
Title: A Phase II Study of Neo-Adjuvant Statin Therapy in Postmenopausal Primary Breast Cancer: A Window-of-Opportunity Study
Brief Title: Study of Statin as Neo-Adjuvant Therapy in Postmenopausal Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lund University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAST1; EudraCT number: 2008-005863-32
Record Dates: First submitted 2008-12-30; First posted 2009-01-01 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-03

CONDITIONS: Breast Cancer; Postmenopausal
Keywords: Breast cancer; Postmenopausal; Neo-adjuvant; Tumor proliferation; Statin; Atorvastatin; Ki67; Translational research; Cell cycle regulators; Gene expression; Genomic profiling; Apoptosis; Window-of-opportunity
MeSH Terms: conditions — Breast Neoplasms | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atorvastatin (Experimental)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin 80 mg daily for two weeks, ending at the day of operation for breast cancer.

SUMMARY:
The purpose of this study is to monitor:

* Tumor biological alterations following two weeks of neo-adjuvant statin therapy.
* Effects of statins on tumor proliferation.
* Functional studies on the mevalonate pathway.

DETAILED DESCRIPTION:
Blood samples and three core biopsies are taken after diagnosis. Treatment with atorvastatin at a daily dosis of 80 mg is initiated 14 days before planned surgery. Translational research will be performed from the core biopsy and blood samples taken before surgery and from the specimen from surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women with primary breast cancer who are candidates for radical surgery.
* Breast tumours clinically ≥ 15 mm, Nx, M0.
* Breast tumours identified on mammography and verified on fine needle aspiration.
* Age > 18 years.
* Performance status of ECOG ≤ 1.
* Laboratory requirements at the day of diagnosis (t1-):Prior to inclusion a normal renal (serum creatinine) and hepatic (transaminases) function (within normal limits) estimated in blood samples is required.
* Prior to patient registration, written informed consent must be given according to ICH/GCP, and national/local regulations.
* Negative pregnancy test for pre menopausal women before inclusion in the trial

Exclusion Criteria:

* Ongoing cholesterol lowering therapy (statins, fibrates, ezetimibe).
* Prior breast cancer treatment.
* Current HRT.
* Known liver disease.
* History of hemorrhagic stroke.
* Psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; these conditions will be discussed with the patient before registration in the trial.
* History of allergic reactions attributed to compounds of similar chemical or biological composition to atorvastatin.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Tumor biological alterations following two weeks of neo-adjuvant statin therapy in postmenopausal breast cancer patients; to evaluate the tumor proliferation using Ki67 as proliferation marker. | After two weeks of treatment with statin therapy.

SECONDARY OUTCOMES:
Assessments of apoptosis using immunohistochemistry. | After two weeks of treatment with statin therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Rose, MD, Principal Investigator — University Hospital Lund
Locations (1):
- University Hospital, Department of Oncology, Lund, Sweden

REFERENCES:
- [Derived] Feldt M, Menard J, Rosendahl AH, Lettiero B, Bendahl PO, Belting M, Borgquist S. The effect of statin treatment on intratumoral cholesterol levels and LDL receptor expression: a window-of-opportunity breast cancer trial. Cancer Metab. 2020 Nov 23;8(1):25. doi: 10.1186/s40170-020-00231-8. PMID 33292612
- [Derived] Feldt M, Bjarnadottir O, Kimbung S, Jirstrom K, Bendahl PO, Veerla S, Grabau D, Hedenfalk I, Borgquist S. Statin-induced anti-proliferative effects via cyclin D1 and p27 in a window-of-opportunity breast cancer trial. J Transl Med. 2015 Apr 29;13:133. doi: 10.1186/s12967-015-0486-0. PMID 25925673